CLINICAL TRIAL: NCT04181697
Title: The HemFitBit-study: Defining Normal Physical Activity in Haemophilia A
Brief Title: HemFitBit, an Observational Study of Physical Activity in People With Moderate and Severe Haemophilia A
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Pål Andre Holme, MD, PhD, Professor of Haematology, Oslo University Hospital
Other Study IDs: 2019/549
Record Dates: First submitted 2019-11-25; First posted 2019-11-29 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Hemophilia A Without Inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PwH A: People with Haemophilia (PwH) A, moderate or severe.
  Interventions: Device: PA measurement with Fitbit Charge 3; Device: PA measurement with Fitbit and ActiGraph GT3X
- Controls: Demographically and seasonally matched non-haemophilia controls.
  Interventions: Device: PA measurement with Fitbit Charge 3

INTERVENTIONS:
Device: PA measurement with Fitbit Charge 3 — Measurement of PA with Fitbit for all participants and controls.
Device: PA measurement with Fitbit and ActiGraph GT3X — Measurement of PA with ActiGraph for a subgroup of 20 participants.
  Groups: PwH A

SUMMARY:
The study aims to describe physical activity (PA) levels in young people with haemophilia A in Norway compared with non-haemophilia controls, and to identify factors influencing PA. This will be conducted through an observational study measuring PA over 12 weeks. Forty young people with moderate and severe haemophilia A will be enrolled. PA data will be compared to demographically and seasonally matched non-haemophilia controls. PA will be measured using the activity tracker Fitbit Charge 3. A subgroup of participants will also wear the hip-worn accelerometer ActiGraph GTX+BT for seven consecutive days in order to validate the two devices against each other.

ELIGIBILITY:
Inclusion Criteria:

* moderate or severe haemophilia A
* no inhibitor
* on continuous prophylaxis

Exclusion Criteria:

* current inhibitor

Ages: 13 Years to 30 Years | Sex: Male
Age Groups: Child, Adult
Study Population: Young people with moderate and severe haemophilia A, without inhibitors and on continuous prophylaxis will be identified from the national registry of PwH.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Physical Activity (PA) volume | 9 months
  PA volume in different intensities
Fulfilment of PA recommendations | 9 months
  Fulfilment of international PA recommendations
Trend in PA over time | 9 months
  Trend in PA and sedentary time over the study period
Physical activity types | 9 months
  Self reported types of PA

SECONDARY OUTCOMES:
Impact of haemophilia on daily life | 9 months
  Work and Classroom Productivity and Activity Impairment (WPAI+CIQ:HS)
Health Related Quality of Life | 9 months
  EuroQol 5Domains 3Levels (EQ-5D-3L) Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension using a three-level scale, and evaluate their overall health status using a Visual analogue scale (VAS) where the bottom rate (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine".
Joint score | 9 months
  Hemophilia Joint Health Score (HJHS 2.1) The Hemophilia Joint Health Score (HJHS) is a validated outcome tool developed for the assessment of joint health in people with hemophilia. The ordinal joint score assesses 9 items in 6 index joints (elbows, knees and ankles). It assesses swelling, duration of swelling, muscle atrophy, crepitus of motion, range of motion (extension and flexion loss), joint pain, strength, and gait. The summation of the 9 HJHS items in 6 index joints provides users with a relative indicator of joint health, with a lower HJHS representing superior joint health.
Ultrasound joint score | 9 months
  Hemophilia Early Arthropathy Detection using Ultrasound (HEAD-US) The ultrasound protocal evaluates the six joints most typically affected in PwH: the elbows, knees, and ankles, in one single examination, providing information about synovium, cartilage, and subchondral bone. Scores for each joint can range between 0 and 8, with higher scores indicating more severe abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No